CLINICAL TRIAL: NCT00952783
Title: A 12 Month, Long-term Follow-up Study of Patients With Actinic Keratosis on Non-head Areas (Trunk and Extremities) Who Have Completed Day 57 in Study PEP005-020
Brief Title: A Long Term Follow up Study of Patients Who Have Completed the PEP005-020 Study
Status: Completed | Type: Observational
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP005-031
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Lesion count

INTERVENTIONS:
Drug: Lesion count — Lesion count in area treated by study drug in a prior study over a 12 month period No drug will be applied during this long-term follow up study. Drug was applied during the primary study.
  Other Names: AK lesion recurrence

SUMMARY:
This study is designed to follow up patients, who have achieved complete clearance of AK lesions (lesion count of 0) at Day 57 in the PEP005-020 study, over a 12 month period to assess both recurrence of Actinic Keratosis (AK) lesions and long term safety in the selected treatment area.

ELIGIBILITY:
Inclusion

* Patient has provided informed consent documented by signing the Informed Consent Form (ICF) prior to any study-related procedures
* Patient achieved complete clearance of AK lesions (lesion count of 0) in the selected treatment area at the Day 57 visit in study PEP005-020

Exclusion

* Concurrent participation in another research study which would involve the selected treatment area (except for any post-study follow-up visits for previous Peplin AK study)
* Early termination from study PEP005-020

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have achieved complete clearance of AK lesions (lesion count of 0) at Day 57 in study PEP005-020
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Summarize treatment area recurrence of AK lesions in the selected treatment area | 12 months

SECONDARY OUTCOMES:
Summarize long-term safety data (incidence of adverse events in the treatment area) | 12 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - Park Avenue Dermatology, Orange Park, Florida
  - Medaphase Inc, Newnan, Georgia
  - Gwinnett Clinical Research Centre, Snellville, Georgia
  - Michigan Center for Research Corp, Clinton Twp, Michigan
  - Henry Ford Health Systems, Detroit, Michigan
  - Dermatology Associates of Rochester, Rochester, New York
  - Oregon Health and Science University, Portland, Oregon
  - Dermatology Research Associates, Nashville, Tennessee
- Australia (3):
  - Dematology on Ward, Adelaide, South Australia
  - Dermatology Institute of Victoria, Melbourne, Victoria
  - St John of God Dermatology, Subiaco, Western Australia

REFERENCES:
- [Derived] Lebwohl M, Shumack S, Stein Gold L, Melgaard A, Larsson T, Tyring SK. Long-term follow-up study of ingenol mebutate gel for the treatment of actinic keratoses. JAMA Dermatol. 2013 Jun;149(6):666-70. doi: 10.1001/jamadermatol.2013.2766. PMID 23553119
- See also: Food and Drug Authority — http://www.fda.gov
- See also: Therapeutic Goods Administration — http://tga.gov.au